CLINICAL TRIAL: NCT03967834
Title: Multimodal Immune Characterization of RAre Soft Tissue Sarcoma - MIRAS Project From SARRA (SARcome RAre) Project of the French Sarcoma Group
Acronym: MIRAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19 SARC 04
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma; Clear Cell Sarcoma; Epithelioid Sarcoma; Perivascular Epithelioid Cell Neoplasms; Desmoplastic Small Round Cell Tumor; Malignant Solitary Fibrous Tumors; Alveolar Soft Part Sarcoma; Epithelioid Hemangioendothelioma; Low Grade Fibromyxoid Sarcoma; Sclerosing Epithelioid Fibrosarcoma
Keywords: Soft Tissue Sarcoma; Clear Cell Sarcoma; Epithelioid Sarcoma; Perivascular Epithelioid Cell Neoplasms; Desmoplastic Small Round Cell Tumor; Malignant Solitary Fibrous Tumors; Alveolar Soft Part Sarcoma; Epithelioid Hemangioendothelioma; Low Grade Fibromyxoid Sarcoma; Sclerosing Epithelioid Fibrosarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Clear Cell; Perivascular Epithelioid Cell Neoplasms; Desmoplastic Small Round Cell Tumor; Sarcoma, Alveolar Soft Part; Hemangioendothelioma, Epithelioid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Soft Tissue Sarcoma (Prospective cohort) (Other)
  Interventions: Other: Patient with Soft Tissue Sarcoma

INTERVENTIONS:
Other: Patient with Soft Tissue Sarcoma — * Tumor specimens will be collected for the study at diagnosis.
  * A blood sample will be collected in all included patients at baseline, after the completion of the treatment (for patients included with a localized disease) or at the time of the first tumoral evaluation (for patients included with a metastatic disease), and at the time of progression.
  * Patient's data (clinical, biological and disease data) will also be collected at baseline visit and then at each time point planned in the center for clinical benefit assessment (i.e. every 2 or 3 months) until progression or for a maximum duration of 5 years.

SUMMARY:
This trial is a translational, open-label, multi-sites, prospective and retrospective cohort study of 500 patients aimed at clinical and biological characterization of sarcoma of rare subtype.

400 patients will be included in this prospective cohort study; they will be identified in the investigating centers in the context of either routine care or a clinical study protocol.

Retrospective cases of patients (100 cases in total) will be identified in all centers through the GSF/GETO clinical databases already setted up (including the clinical base Conticabase).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Diagnosis of one of the following rare sarcoma subtype, confirmed by RRePS network:

   * Clear Cell Sarcoma (CCS)
   * Epithelioid Sarcoma (ES)
   * Perivascular Epithelioid Cell neoplasm (PEComa)
   * Desmoplastic Small Round Cell Tumours (DSRCT)
   * Malignant Solitary Fibrous Tumours (mSFT)
   * Alveolar Soft Part Sarcoma (ASPS)
   * Epithelioid Hemangioendothelioma (EH)
   * Low-Grade Fibromyxoid Sarcoma (LGFS)
   * Sclerosing Epithelioid Fibrosarcoma (SEF).
3. Localized/locally advanced or metastatic disease.
4. In case of localized disease, treatment must not have been yet initiated before inclusion (except surgical excision).
5. In case of metastatic disease, project of new line of systemic treatment must have been decided before inclusion.
6. Patient followed in the center within a standard of care procedure or clinical trial.
7. Archived tumor specimen at initial diagnosis available (before treatment initiation).
8. Evaluable disease (measurable as per RECIST 1.1) or not.
9. ECOG Performance status 0-3.
10. Patient able to participate and willing to give informed consent prior to performance of any study-related procedures.
11. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Diagnosis of all other histotypes of soft tissue sarcoma.
2. Any condition contraindicated with procedures required by the protocol.
3. Known history of positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
5. Pregnant or breast-feeding woman.
6. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival for patients with localized disease. | 60 months for each patients
Progression-free survival for patients with metastatic disease. | 60 months for each patients

SECONDARY OUTCOMES:
Cancer-Testis Antigens (CTA) expression. | 60 months for each patients
The rate of patients presenting high-risk CINSARC (Complexity Index in SARComas) signature. | 60 months for each patients
Overall survival. | 60 months for each patients

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Chu Besancon - Site Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Chu Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Chu de Marseille - Hopital de La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin - Site Port-Royal, Paris
  - Institut Curie, Paris
  - Chu Poitiers, Poitiers
  - Institut Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de L'Ouest - Site Rene Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif